CLINICAL TRIAL: NCT06523010
Title: The Effect of Talocrural Joint Manipulation on Static Balance in Patients With Stroke
Brief Title: Talocrural Joint Manipulation in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BEUFTR-5
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: postural balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The patients enrolled in the study will receive placebo talocrural joint traction and talocrural joint traction in a randomized sequence. The order of the interventions will be determined by flipping a coin.
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluator and the researcher administering the intervention will be different. The interventions will be administered to participants randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Talocrural Joint Manipulation Group (Placebo Comparator): Each group will receive both placebo and real talocrural joint manipulations in a randomized cross-over design. There will be a minimum interval of 48 hours between the interventions. Data obtained after the real manipulation will be recorded as the placebo comparator group data.
  Interventions: Other: Talocrural Joint Manipulation; Other: Placebo Talocrural Joint Manipulation
- Talocrural Joint Manipulation Group (Active Comparator): Each group will receive both placebo and real talocrural joint manipulations in a randomized cross-over design. There will be a minimum interval of 48 hours between the interventions. Data obtained after the real manipulation will be recorded as the active comparison group data.
  Interventions: Other: Talocrural Joint Manipulation; Other: Placebo Talocrural Joint Manipulation

INTERVENTIONS:
Other: Talocrural Joint Manipulation — This technique, aiming to increase ankle dorsiflexion and mechanoreceptor activation, is based on the application of high velocity low amplitude traction to the joint.
Other: Placebo Talocrural Joint Manipulation — This intervention is a classic method used to evaluate the effect of talocrural joint manipulation.

SUMMARY:
The primary aim of the study is to investigate the effect of talocrural joint manipulation on the static balance of patients with stroke. The secondary aim of this study is to investigate the effect of talocrural joint manipulation on the dorsiflexion range of motion of patients with stroke.

DETAILED DESCRIPTION:
The study, utilizing a randomized crossover design, is planned to be conducted on a minimum of 26 patients with stroke who meet the inclusion and exclusion criteria. Patients included in the study will be randomly assigned to receive both placebo talocrural joint manipulation and talocrural joint manipulation treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Two months or longer elapsed since the stroke,
* 2. A Mini-Mental State Examination score of 24 or higher,
* 3. The ability to stand independently for 20 seconds or more,
* 4. The ability to walk independently for 10 meters with the use of walking aids or orthoses if necessary,
* 5. Being between 45 and 75 years of age,
* 6. Having a Brunnstrom stage of 4 or above

Exclusion Criteria:

* 1. The presence of severe osteoarthritis in the lower extremity,
* 2. The presence of cancer or diabetic neuropathy,
* 3. The presence of vestibular disorder,
* 4. The presence of lower extremity ulceration or amputation,
* 5. History of vertigo,
* 6. Alcohol consumption within the last 24 hours,
* 7. Hemodynamic instability,
* 8. Diagnosis of posterior circulation stroke involving the basilar artery and cerebellum,
* 9. The presence of other neurological disorders (such as multiple sclerosis, Parkinson's disease),
* 10. Having experienced an acute lower extremity injury in the last six weeks,
* 11. History of lower extremity surgery

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ömer dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; burak mavuş, Mr., Principal Investigator — Bolu Abant İzzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital
Locations (1):
- Bolu İzzet Baysal Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Bolu, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Tyson SF, Hanley M, Chillala J, Selley A, Tallis RC. Balance disability after stroke. Phys Ther. 2006 Jan;86(1):30-8. doi: 10.1093/ptj/86.1.30. PMID 16386060
- [Background] Yates JS, Lai SM, Duncan PW, Studenski S. Falls in community-dwelling stroke survivors: an accumulated impairments model. J Rehabil Res Dev. 2002 May-Jun;39(3):385-94. PMID 12173758
- [Background] Divani AA, Vazquez G, Barrett AM, Asadollahi M, Luft AR. Risk factors associated with injury attributable to falling among elderly population with history of stroke. Stroke. 2009 Oct;40(10):3286-92. doi: 10.1161/STROKEAHA.109.559195. Epub 2009 Jul 23. PMID 19628798
- [Background] Lamb SE, Ferrucci L, Volapto S, Fried LP, Guralnik JM; Women's Health and Aging Study. Risk factors for falling in home-dwelling older women with stroke: the Women's Health and Aging Study. Stroke. 2003 Feb;34(2):494-501. PMID 12574566
- [Background] Powden CJ, Hogan KK, Wikstrom EA, Hoch MC. The Effect of 2 Forms of Talocrural Joint Traction on Dorsiflexion Range of Motion and Postural Control in Those With Chronic Ankle Instability. J Sport Rehabil. 2017 May;26(3):239-244. doi: 10.1123/jsr.2015-0152. Epub 2016 Aug 24. PMID 27632835
- [Background] Hoch MC, Andreatta RD, Mullineaux DR, English RA, Medina McKeon JM, Mattacola CG, McKeon PO. Two-week joint mobilization intervention improves self-reported function, range of motion, and dynamic balance in those with chronic ankle instability. J Orthop Res. 2012 Nov;30(11):1798-804. doi: 10.1002/jor.22150. Epub 2012 May 18. PMID 22610971
- [Background] Hoch MC, McKeon PO. Joint mobilization improves spatiotemporal postural control and range of motion in those with chronic ankle instability. J Orthop Res. 2011 Mar;29(3):326-32. doi: 10.1002/jor.21256. Epub 2010 Sep 30. PMID 20886654
- [Background] Alamer A, Melese H, Getie K, Deme S, Tsega M, Ayhualem S, Birhanie G, Abich Y, Yitayeh Gelaw A. Effect of Ankle Joint Mobilization with Movement on Range of Motion, Balance and Gait Function in Chronic Stroke Survivors: Systematic Review of Randomized Controlled Trials. Degener Neurol Neuromuscul Dis. 2021 Sep 1;11:51-60. doi: 10.2147/DNND.S317865. eCollection 2021. PMID 34512072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in compliance with the principles outlined in the 1964 Declaration of Helsinki, and it took place at İzzet Baysal Physical Therapy and Rehabilitation Training and Research Hospital between August 2024, and December 2024.
Pre-assignment Details: Before group allocation, one individual was excluded from the study due to being over 75 years of age, 29 individuals due to cognitive dysfunction, 2 individuals due to lower extremity amputation, and 90 individuals because their Brunnstrom recovery stage was below stage four.
Groups:
- Placebo Talocrural Joint Manipulation Group: Patients in this group will first receive a placebo talocrural joint manipulation, followed by the actual talocrural joint manipulation after a washout period of at least 48 hours.
- Talocrural Joint Manipulation Group: Patients in this group will first receive the actual talocrural joint manipulation, followed by the placebo talocrural joint manipulation after a washout period of at least 48 hours.
Period: Overall Study
Arm/Group | Placebo Talocrural Joint Manipulation Group | Talocrural Joint Manipulation Group
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants were involved in the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.21 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.36 (2.99)
Height [Mean (Standard Deviation); unit: centimeter] | 166.84 (9.29)
Weight [Mean (Standard Deviation); unit: kilogram] | 78.93 (6.74)

OUTCOME MEASURES:

1. Primary Outcome: Overall Stability Index Measurement
Description: Overall stability index, evaluated using the Biodex Balance System. Overall stability index scores were derived from calculations of deviations from the center of gravity in the anteroposterior and mediolateral axes by the device. A lower score indicates smaller deviation and better postural stability. The assessment was conducted on a stable platform with three 20-second repetitions interspersed with 10-second rest periods. Participants remained standing during the rest periods, and the device automatically computed the average of the three repetitions. As the general stability index value increases, overall stability decreases. No definable minimum or maximum theoretical value.
Time Frame: Change from baseline overall stability immediately after intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Placebo Only: Only the pre- and post-intervention values of the patients in this group who received placebo manipulation were taken into account.
- Talocrural Manipulation Only: Only the pre- and post-intervention values of the patients in this group who received real manipulation were taken into account.
Arm/Group | Placebo Only | Talocrural Manipulation Only
Number analyzed (Participants) | 64 | 64
units on a scale | 17.5 [8 to 28] | 9 [2 to 22]

2. Secondary Outcome: Mediolateral Stability Index Measurement
Description: Mediolateral stability index, evaluated using the Biodex Balance System. Mediolateral stability index scores were derived from calculations of deviations from the center of gravity in the mediolateral axis by the device. As the mediolateral index value increases, mediolateral stability decreases. No definable minimum or maximum theoretical value.
Time Frame: Change from baseline mediolateral stability immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Only | Talocrural Manipulation Only
Number analyzed (Participants) | 64 | 64
units on a scale | 6.96 (2.59) | 4.87 (2.76)

3. Secondary Outcome: Anteroposterior Stability Index Measurement
Description: Anteroposterior stability index, evaluated using the Biodex Balance System. Anteroposterior stability index scores were derived from calculations of deviations from the center of gravity in the anteroposterior axis by the device. As the overall anteroposterior stability value increases, anteroposterior stability decreases. No definable minimum or maximum theoretical value.
Time Frame: Change from baseline anteroposterior stability immediately after intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Only | Talocrural Manipulation Only
Number analyzed (Participants) | 64 | 64
units on a scale | 10 [4 to 14] | 5.5 [1 to 12]

4. Secondary Outcome: Ankle Dorsiflexion Range of Motion Measurement With Knee in Extended and Flexed Positions
Description: The patient was asked to stand facing the wall and place their hands on the wall at shoulder width apart, with the affected foot positioned behind and the knee in full extension. Then, without lifting the back foot or compromising knee extension, the patient was instructed to reach forward as far as possible. Subsequently, the calcaneal tubercle was placed one centimeter above the floor, and the measurement was taken with a water level gauge attached to the phone. The same measurement was repeated with the knee in flexion (20 degrees or more).
Time Frame: Change from baseline ankle dorsiflexion range of motion immediately after intervention
Measure: Median (Inter-Quartile Range); unit: average of ankle dorsi flexion degree
Arm/Group | Placebo Only | Talocrural Manipulation Only
Number analyzed (Participants) | 64 | 64
average of ankle dorsi flexion degree
  Knee flexed dorsi flexion | 13 [8 to 35] | 22.5 [11 to 39]
  Knee extended dorsi flexion | 10 [7 to 27] | 18.5 [7 to 36]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of one week
Groups:
- All Participants in the Study: All study participants were involved in the study.
Arm/Group | All Participants in the Study
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

LIMITATIONS AND CAVEATS:
The study has some limitations. Firstly, due to the short follow-up period, the medium-and long-term effects of talocrural joint manipulation on postural stability and ankle mobility could not be evaluated. For this reason, further studies are needed to determine the medium- and long-term effects. Secondly, since accessory joint movements were not evaluated, no conclusions could be drawn regarding the effect of talocrural joint manipulation on accessory joint movements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT06523010/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT06523010/SAP_001.pdf